CLINICAL TRIAL: NCT02193269
Title: Cognitive Effects of Minocycline in Humans
Brief Title: The Effects of Minocycline in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Mehmet Sofuoglu, M.D.,Ph.D., Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1304011871
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Memory Impairment
Keywords: Abstinent cocaine users; minocycline; antibiotic
MeSH Terms: conditions — Memory Disorders; cyclopia sequence | interventions — Sugars; Minocycline; Tetracycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator): 0.0mg
  Interventions: Drug: Minocycline
- Minocycline (Active Comparator): 200mg
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Sugar pill — you will receive 0.0 mg as a single daily dose for 4 days
  Other Names: sugar pill, placebo
  Arms: Minocycline
Drug: Minocycline — you will receive 200 mg as a single daily dose for 4 days
  Other Names: tetracycline antibiotic
  Arms: sugar pill

SUMMARY:
To determine minocycline's effects on cognitive performance and measures of mood in abstinent cocaine users. Minocycline is a tetracycline derivative antibiotic that also inhibits microglia activation and the release of pro-inflammatory cytokines, chemokines, and nitric oxide (NO) production. Previous animal and human studies suggest that minocycline may have utility as a treatment for cocaine addiction.

DETAILED DESCRIPTION:
We are proposing a randomized, double-blind, crossover study. A total of 40 male and or female subject completers will have two 4-day treatment periods, in which they will be randomized to minocycline (200 mg/day) or placebo. During the first 3 days of each treatment period, subjects will have daily clinic visits for medication administration and monitoring of adverse events. On Day 4, subjects will have an experimental session in which measures of mood and cognitive performance will be obtained. Following a washout period, ranging from 5 to 15 days, subjects will be crossed over to the alternative treatment.

This study began July 2013; currently 7 subjects were randomized with 5 completers and two drop outs. This study is in data analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, between the ages of 21 and 50 who fulfill criteria for past cocaine dependence according to DSM-IV criteria;
* No cocaine use for the past 30 days;
* No other current dependence or abuse of other drugs of abuse or alcohol (except cocaine and tobacco);
* No current medical problems and normal ECG;
* For women, not pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* current major psychiatric illnesses including mood, psychotic, or anxiety disorders;
* history of major medical illnesses; including liver diseases, heart disease, or other medical conditions that the physician investigator deems contraindicated for the subject to be in the study
* Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants) or drugs that would be expected to have major interactions with drugs to be tested, e.g., benzodiazepines, codeine, percocet, and other opiate drugs that will interact with methadone.
* Liver function tests (ALT or AST) greater than 3 times normal.
* Allergy to minocycline or other tetracyclines.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Rapid Visual information Processing | 2 yrs
  Cognitive Test to determine the speed of Visual information

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Veteran Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No